CLINICAL TRIAL: NCT03357341
Title: Enabling Innovative Respiratory Real World Evidence Generation: Sensor and EHR Integration Pilot Study
Brief Title: Sensor and Electronic Health Records (EHR) Integration Pilot Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Geisinger HealthPlan (Industry)
Responsible Party: Sponsor
Other Study IDs: 207223; HO-17-17827 (Other: Track HO identifier)
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: electronic health record; Pilot; COPD; Sensor; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Albuterol; Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- COPD cohort: Approximately 100 subjects with COPD identified through integrated EHR records will be enrolled.
  Interventions: Device: Mobile spirometer; Device: Device sensor; Drug: Salbutamol; Device: Activity monitor; Other: electronic diary card; Other: CAT
- Asthma cohort: Approximately 100 subjects with asthma identified through integrated EHR records will be enrolled.
  Interventions: Device: Mobile spirometer; Device: Device sensor; Drug: Salbutamol; Device: Activity monitor; Other: ACT

INTERVENTIONS:
Device: Mobile spirometer — Mobile spirometer will be used to measure FEV1 values weekly.
Device: Device sensor — Sensors will be attached to rescue and maintenance inhalers to measure use of rescue medication and maintenance therapy.
Drug: Salbutamol — Salbutamol MDI will be given as a rescue medication to be used on an as needed basis in this study.
Device: Activity monitor — Subjects will be required to wear activity monitors daily to record their physical activity.
Other: electronic diary card — Electronic diary card will be completed daily by subjects in COPD cohort.
  Groups: COPD cohort
Other: CAT — Subjects will be required to complete CAT monthly.
  Groups: COPD cohort
Other: ACT — Subjects will be required to complete ACT monthly.
  Groups: Asthma cohort

SUMMARY:
This is a pilot study that will evaluate the feasibility of collecting increasing amounts of clinical study data from subjects through sensor and web/app based methods and integrating it with data from their EHR to facilitate more efficient and meaningful research with acceptable quality. Approximately 100 subjects with asthma and 100 subjects with chronic obstructive pulmonary disease (COPD) will be enrolled in this prospective study. The subjects will be identified through integrated EHR records following which eligible subjects will receive study devices and training on proper use of the devices at Baseline visit. Data will be collected remotely from subject reports, devices and sensors over six months.

ELIGIBILITY:
Inclusion Criteria:

COPD cohort

* Provide signed and dated informed consent form.
* Be willing to comply with all study procedures and be available for the duration of the study.
* Age >=40 years
* Diagnosed with COPD, defined as COPD listed on the subject's problem list and one of the following: a) At least one inpatient hospitalization with a COPD diagnosis listed as the primary or secondary diagnosis (J41.x, J42.x, J44.x [chronic bronchitis], J43.9 [emphysema] or J44.9 [Chronic obstructive pulmonary disease, unspecified]) in the last 12 months b) At least two outpatient encounters with a diagnosis of COPD exacerbation (J44.1), Acute bronchitis (J20.x), or bronchitis (J40) listed as the primary or secondary diagnosis, with different dates of service in the last 12 months c) At least one emergency room encounter with a COPD diagnosis (J41.x, J42.x, J44.x, J43.9, J44.9) listed as the primary or secondary diagnosis in the last 12 months d) At least two urgent care encounters with different dates of service, with a COPD diagnosis (J41.x, J42.x, J44.x, J43.9, J44.9) listed as the primary or secondary diagnosis in the last 12 months.
* At least one order for an inhaled COPD medication during the prior year.
* More than 12 months of data available in the integrated EHR data prior to date of screening.

Asthma cohort

* Provide signed and dated informed consent form.
* Be willing to comply with all study procedures and be available for the duration of the study.
* Age >=18 years
* Diagnosed with asthma, defined as asthma listed on the subject's problem list and one of the following: a) At least one inpatient hospitalization with an asthma diagnosis (J45.x) listed as the primary or secondary diagnosis in the last 12 months. b) At least one emergency room encounter with an asthma diagnosis (J45.x) listed as the primary or secondary diagnosis in the last 12 months c) at least two urgent care encounters, with different dates of service, with an asthma diagnosis (J45.x) listed as the primary or secondary diagnosis in the last 12 months d) At least three or more prescriptions or prescription refills in the past 12 months for any combination of the following: an inhaled glucocorticoid with or without a second controller (Montelukast, Theophylline, a long-acting beta agonist [LABA] alone) or a combination drug with a LABA and an inhaled glucocorticoid.
* More than 12 months of data available in the integrated EHR data prior to date of screening.

Exclusion Criteria:

COPD cohort

* Inability/Unwillingness to use the required devices, or
* Inability to read and understand English Asthma cohort
* Inability/Unwillingness to use the required devices
* Inability to read and understand English
* Diagnosis of COPD listed on problem list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two cohorts consisting of approximately 100 subjects each with COPD and asthma identified through EHR database analyses will be included.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Danville, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective observational study that included two cohorts of participants identified through electronic health records (EHR) within the Geisinger Health System (GHS) database. The study was conducted at a single center in the United States.
Pre-assignment Details: A total of 194 participants were enrolled and followed up for six months. The study data was captured remotely via sensors and devices provided by GlaxoSmithKline (GSK) to the participants, or via extraction of EHR data.
Groups:
- Asthma Cohort: Asthma participants were identified via EHR database analyses, study provider referral (asthma diagnoses with and without specialist confirmation) or recruited from sites of usual care. Participants attended two visits at the Baseline (Visit 1) and approximately six months later (Visit 2). At Visit 2, the participants returned the study devices and attended exit interview to provide relevant feedback.
- COPD Cohort: Participants with chronic obstructive pulmonary disease (COPD) were identified via EHR database analyses, study provider referral (COPD diagnoses with and without specialist confirmation) or recruited from sites of usual care. Participants attended two visits at the Baseline (Visit 1) and approximately six months later (Visit 2). At Visit 2, the participants returned the study devices and attended exit interview to provide relevant feedback.
Period: Overall Study
Arm/Group | Asthma Cohort | COPD Cohort
Started | 96 | 98
Completed | 89 | 86
Not Completed | 7 | 12
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 4 | 5
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthma Cohort | COPD Cohort | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 59 [44 to 67] | 64 [57 to 71] | 62 [52 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 66 | 129
  Male | 33 | 32 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 93 | 94 | 187
  African-American | 1 | 4 | 5
  South East Asian | 1 | 0 | 1
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 is an important measure of pulmonary function and is the maximum amount of air that can be forced out in one second after taking a deep breath. FEV1 was measured using spirometry. Participants were given a hand-held spirometer with instructions on its proper use. Baseline (Week 1) measurement was taken in clinic and the participants were instructed to perform home spirometry on a weekly basis for the remainder of the study. The spirometry use was linked to the Propeller Health application on the iPad, which provided visual cues for the spirometry and sent the data to the central database after completion of the session. Change from Baseline was calculated as the value at specified time point minus Baseline value. Change from Baseline in FEV1 at 4-weekly intervals is presented.
Time Frame: Baseline (Week 1) and Weeks 5, 9, 13, 17, 21 and 25
Population: All Enrolled Population: Includes participants with asthma and COPD identified via EHR database. Total of 73 and 68 participants were included in the analysis; however only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Median (Inter-Quartile Range); unit: Liter
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 73 | 68
Liter
  Week 5, n=61, 44: number analyzed (Participants) | 61 | 44
  Week 5, n=61, 44 | -0.03 [-0.23 to 0.14] | 0.07 [-0.08 to 0.17]
  Week 9, n=61,39: number analyzed (Participants) | 61 | 39
  Week 9, n=61,39 | -0.09 [-0.28 to 0.11] | -0.08 [-0.26 to 0.03]
  Week 13, n=57, 40: number analyzed (Participants) | 57 | 40
  Week 13, n=57, 40 | -0.06 [-0.22 to 0.14] | -0.10 [-0.22 to 0.06]
  Week 17, n=54, 38: number analyzed (Participants) | 54 | 38
  Week 17, n=54, 38 | -0.11 [-0.27 to 0.05] | -0.15 [-0.23 to 0.09]
  Week 21, n=33, 28: number analyzed (Participants) | 33 | 28
  Week 21, n=33, 28 | -0.07 [-0.22 to 0.08] | -0.19 [-0.51 to 0.00]
  Week 25, n=26, 14: number analyzed (Participants) | 26 | 14
  Week 25, n=26, 14 | -0.12 [-0.24 to 0.18] | -0.10 [-0.27 to 0.01]

2. Primary Outcome: Median Number of Steps Per Day
Description: The physical activity was captured using a waist-worn accelerometer. A valid day was defined as a day where the activity monitor detected that it was worn for at least 8 hours during that day. Data for three or more valid days were required to generate data for weekly step counts.
Time Frame: Weeks 1, 5, 9, 13, 17, 21 and 25
Population: All Enrolled Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Median (Inter-Quartile Range); unit: Steps per day
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 72 | 68
Steps per day
  Week 1, n=72, 68 | 3574 [2321 to 5584] | 2186 [1185 to 3320]
  Week 5, n=53, 54: number analyzed (Participants) | 53 | 54
  Week 5, n=53, 54 | 4547 [1956 to 6021] | 2446 [1281 to 3832]
  Week 9, n=52,42: number analyzed (Participants) | 52 | 42
  Week 9, n=52,42 | 3270 [2161 to 6358] | 2312 [1335 to 3605]
  Week 13, n=52, 42: number analyzed (Participants) | 52 | 42
  Week 13, n=52, 42 | 3124 [1944 to 6425] | 2117 [1150 to 3390]
  Week 17, n=47, 37: number analyzed (Participants) | 47 | 37
  Week 17, n=47, 37 | 3962 [2160 to 6637] | 1583 [1148 to 2752]
  Week 21, n=34, 31: number analyzed (Participants) | 34 | 31
  Week 21, n=34, 31 | 3816 [1498 to 6547] | 1702 [912 to 3645]
  Week 25, n=23, 20: number analyzed (Participants) | 23 | 20
  Week 25, n=23, 20 | 3431 [1822 to 6501] | 2239 [1012 to 3139]

3. Primary Outcome: Median Daily Activity Level Based on Vector Magnitude Counts.
Description: The physical activity was captured using a waist-worn accelerometer. Vector magnitude in counts are accelerations in 3 dimensions that indicate activity. More counts is associated with more activity.
Time Frame: Weeks 1, 5, 9, 13, 17, 21 and 25
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Vector magnitude counts
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 72 | 68
Vector magnitude counts
  Week 1, n=72, 68 | 512 [407 to 658] | 378 [288 to 492]
  Week 5, n=53, 54: number analyzed (Participants) | 53 | 54
  Week 5, n=53, 54 | 475 [375 to 669] | 415 [302 to 578]
  Week 9, n=52, 42: number analyzed (Participants) | 52 | 42
  Week 9, n=52, 42 | 483 [348 to 629] | 389 [290 to 523]
  Week 13, n=52, 42: number analyzed (Participants) | 52 | 42
  Week 13, n=52, 42 | 469 [342 to 685] | 384 [268 to 541]
  Week 17, n=47, 37: number analyzed (Participants) | 47 | 37
  Week 17, n=47, 37 | 490 [375 to 670] | 342 [272 to 434]
  Week 21, n=34, 31: number analyzed (Participants) | 34 | 31
  Week 21, n=34, 31 | 525 [359 to 683] | 359 [242 to 608]
  Week 25, n=23, 20: number analyzed (Participants) | 23 | 20
  Week 25, n=23, 20 | 446 [343 to 661] | 412 [311 to 648]

4. Primary Outcome: Patient Reported Outcome (PRO) Active Total Score
Description: The PROactive tool is used to investigate dimensions of physical activity (symptoms, distress, difficulties, amount etc.) that are judged as being essential by participants living with COPD. The clinic visit version of PRO was used, and was offered via the participant's electronic PRO application every 28 days. This version of PRO includes 14 items, measuring a physical activity 'Total Score' with 2 domains ('amount' and 'difficulty'). The 'amount' domain is covered by 2 items (amount of walking outside and chores outside) and by 2 activity monitor outputs (vector magnitude units per minute [VMU/min] and steps per day). The 'difficulty' domain is covered by 10 items. Each domain score is based on the simple addition of items (scale ranging from 0 to 15 for amount domain and 0 to 40 for difficulty domain), and then scaled from 0 to 100. 'Total Score' is calculated as the sum of the two domains (amount and difficulty) divided by two, thus scored from 0 (worse) to 100 (much better).
Time Frame: Weeks 2, 6, 10, 14, 18, 22 and 26
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 54 | 58
Scores on a scale
  Week 2, n=54, 58 | 75 [66.5 to 78.5] | 60.3 [54.5 to 69]
  Week 6, n=40, 52: number analyzed (Participants) | 40 | 52
  Week 6, n=40, 52 | 75 [63.8 to 79.3] | 59 [55.3 to 66]
  Week 10, n=35,36: number analyzed (Participants) | 35 | 36
  Week 10, n=35,36 | 73 [63.5 to 78.5] | 62.5 [53.5 to 69.5]
  Week 14, n=36, 36: number analyzed (Participants) | 36 | 36
  Week 14, n=36, 36 | 73.5 [65.5 to 79.3] | 58.5 [49.5 to 68.3]
  Week 18, n=22, 22: number analyzed (Participants) | 22 | 22
  Week 18, n=22, 22 | 75 [70 to 78.5] | 57.5 [52.5 to 61.5]
  Week 22, n=21, 23: number analyzed (Participants) | 21 | 23
  Week 22, n=21, 23 | 76.5 [67 to 81] | 56.5 [48.5 to 63.5]
  Week 26, n=15, 12: number analyzed (Participants) | 15 | 12
  Week 26, n=15, 12 | 75.5 [67 to 79] | 58 [56.3 to 67.8]

5. Primary Outcome: PROactive Amount Domain Score
Description: The PROactive tool is used to investigate dimensions of physical activity (symptoms, distress, difficulties, amount etc.) that are judged as being essential by participants living with COPD. The clinic visit version of the PRO was used in this study, and was offered via the participant's electronic PRO application every 28 days. This version of the PRO includes 14 items, measuring a physical activity 'Total Score' with 2 domains (amount and difficulty). The amount domain is covered by 2 items (amount of walking outside and chores outside) and by 2 activity monitor outputs (vector magnitude units per minute [VMU/min] and steps per day). Amount domain score is based on the simple addition of items (scale ranging from 0 to 15) and then scaled from 0 to 100.
Time Frame: Weeks 2, 6, 10, 14, 18, 22 and 26
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 54 | 58
Scores on a scale
  Week 2, n=54, 58 | 61 [52 to 70] | 52 [48 to 57]
  Week 6, n=40, 52: number analyzed (Participants) | 40 | 52
  Week 6, n=40, 52 | 61 [52 to 65] | 54 [48 to 61]
  Week 10, n=35,36: number analyzed (Participants) | 35 | 36
  Week 10, n=35,36 | 57 [52 to 65] | 57 [48 to 61]
  Week 14, n=36, 36: number analyzed (Participants) | 36 | 36
  Week 14, n=36, 36 | 59 [52 to 70] | 52 [44 to 63]
  Week 18, n=22, 22: number analyzed (Participants) | 22 | 22
  Week 18, n=22, 22 | 61 [57 to 75] | 52 [48 to 61]
  Week 22, n=21, 23: number analyzed (Participants) | 21 | 23
  Week 22, n=21, 23 | 61 [57 to 75] | 52 [39 to 61]
  Week 26, n=15, 12: number analyzed (Participants) | 15 | 12
  Week 26, n=15, 12 | 61 [57 to 70] | 54 [46 to 57]

6. Primary Outcome: PROactive Difficulty Domain Score
Description: The PROactive tool is used to investigate dimensions of physical activity (symptoms, distress, difficulties, amount etc.) that are judged as being essential by participants living with COPD. The clinic visit version of the PRO was used in this study, and was offered via the participant's electronic PRO application every 28 days. This version of the PRO includes 14 items, measuring a physical activity 'Total Score' with 2 domains ('amount' and 'difficulty'). The 'difficulty' domain is covered by 10 items. The difficulty domain score is based on the simple addition of items (0 to 40), which is then scaled from 0 (worse) to 100 (much better).
Time Frame: Weeks 2, 6, 10, 14, 18, 22 and 26
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 68 | 83
Scores on a scale
  Week 2, n=68, 83 | 84.5 [73 to 94] | 66 [60 to 75]
  Week 6, n=57, 77: number analyzed (Participants) | 57 | 77
  Week 6, n=57, 77 | 86 [68 to 94] | 63 [56 to 77]
  Week 10, n=54, 65: number analyzed (Participants) | 54 | 65
  Week 10, n=54, 65 | 82 [72 to 92] | 65 [55 to 73]
  Week 14, n=49, 56: number analyzed (Participants) | 49 | 56
  Week 14, n=49, 56 | 83 [79 to 94] | 66 [56.5 to 83]
  Week 18, n=39, 41: number analyzed (Participants) | 39 | 41
  Week 18, n=39, 41 | 83 [75 to 92] | 61 [56 to 72]
  Week 22, n=47, 50: number analyzed (Participants) | 47 | 50
  Week 22, n=47, 50 | 86 [77 to 92] | 65.5 [53 to 70]
  Week 26, n=28, 37: number analyzed (Participants) | 28 | 37
  Week 26, n=28, 37 | 86 [78 to 94] | 65 [55 to 72]

7. Primary Outcome: Evaluating Respiratory Symptoms (E-RS) in COPD Total Score-COPD Cohort Only
Description: The E-RS: COPD scale is a derivative instrument used to measure the effect of treatment on the severity of respiratory symptoms in stable COPD. The E-RS utilizes the 11 respiratory symptom items contained in the 14-item Exacerbations of Chronic pulmonary disease Tool (EXACT). For the COPD cohort specifically, the daily EXACT was offered each evening. The domains included: respiratory symptoms (RS)-breathlessness (RS-BRL comprised of 5 items, score range [0-17]), RS-cough and sputum (RS-CSP comprised of 3 items, score range [0-11]), and RS-chest symptoms (RS-CSY comprised of 3 items, score range [0-12]). The total score was derived by summing the 11-item scores and ranged between 0-40 with higher values indicating severe respiratory symptoms. Scores for the week were summarized for each COPD participant where they completed the questionnaire on three or more days during the study week
Time Frame: Weeks 1, 5, 9, 13, 17, 21 and 25
Population: All Enrolled Population.Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | COPD Cohort
Number analyzed (Participants) | 72
Scores on a scale
  Week 1, n=72 | 16.5 [11.5 to 22.3]
  Week 5, n=66: number analyzed (Participants) | 66
  Week 5, n=66 | 17.8 [12.0 to 23.5]
  Week 9, n=60: number analyzed (Participants) | 60
  Week 9, n=60 | 17.1 [11.7 to 25.9]
  Week 13, n=56: number analyzed (Participants) | 56
  Week 13, n=56 | 15.5 [12.4 to 23.4]
  Week 17, n=52: number analyzed (Participants) | 52
  Week 17, n=52 | 15.8 [11.9 to 23.8]
  Week 21, n=43: number analyzed (Participants) | 43
  Week 21, n=43 | 16.3 [11.5 to 23.0]
  Week 25, n=41: number analyzed (Participants) | 41
  Week 25, n=41 | 15.3 [10.3 to 21.4]

8. Primary Outcome: Exacerbations of Chronic Pulmonary Disease Tool (EXACT) Event Rate-COPD Cohort Only
Description: EXACT is a 14-item diary that measures respiratory symptoms and function. The total score for EXACT ranges from 0-100, higher scores indicate more severe symptoms. EXACT events are considered worsening of symptom scores above the individual's Baseline value over multiple consecutive days.
Time Frame: Up to 6 months
Population: All Enrolled Population.
Measure: Number; unit: Events per participant per year
Arm/Group | COPD Cohort
Number analyzed (Participants) | 98
Events per participant per year | 2.06

9. Primary Outcome: Number of Primary Care Visits for Asthma Conditions or COPD
Description: The number of primary care visits (including ambulatory, home and phone) for asthma conditions or COPD were summarized using data from EHR-based healthcare utilization.
Time Frame: Up to 6 months
Population: All Enrolled Population.
Measure: Number; unit: Visits
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Visits
  Ambulatory | 23 | 79
  Home | 1 | 21
  Phone | 4 | 17

10. Primary Outcome: Number of Secondary Care Visits for Asthma Conditions or COPD
Description: The number of secondary care visits (that is, inpatient hospitalization and emergency department [ED]) for asthma conditions or COPD were summarized using data from EHR-based healthcare utilization
Time Frame: Up to 6 months
Population: All Enrolled Population
Measure: Number; unit: Visits
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Visits
  Inpatient hospitalization | 0 | 0
  ED visits | 0 | 0

11. Primary Outcome: Number of All Primary Care Visits
Description: The number of all primary care visits (including ambulatory, home and phone) were summarized using data from EHR-based healthcare utilization
Time Frame: Up to 6 months
Population: All Enrolled Population
Measure: Number; unit: Visits
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Visits
  Ambulatory | 426 | 598
  Home | 7 | 55
  Phone | 87 | 116

12. Primary Outcome: Number of All Secondary Care Visits
Description: The number of all secondary care visits (that is, inpatient hospitalization and ED) were summarized using data from EHR-based healthcare utilization
Time Frame: Up to 6 months
Population: All Enrolled Population
Measure: Number; unit: Visits
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Visits
  Inpatient hospitalization | 0 | 0
  ED visits | 0 | 0

13. Primary Outcome: Number of Participants With New Prescriptions
Description: New treatments that were prescribed for respiratory-related conditions (Short-acting beta-agonists [SABA], Inhaled corticosteroid (ICS)/long-acting beta-agonist [LABA] combinations, Oral corticosteroids [OCS], Leukotriene modifiers [LEUK], ICS, Long-acting muscarinic antagonists [LAMA], SABA/short-acting muscarinic antagonist [SAMA] combinations, Anti-cholinergics [a-CHOL], LABA/LAMA, ICS/LABA/LAMA, Phosphodiesterase type 4 inhibitors [PDE4], Anti-immunoglobulin E [a-IgE], LABA, and Interleukin-5 inhibitors [IL-5]) were summarized using data from EHR-based healthcare utilization. Some participants may have received prescriptions in more than one medication category.
Time Frame: Up to 6 months
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Participants
  SABA | 85 | 85
  ICS/LABA | 59 | 48
  OCS | 33 | 52
  LEUK | 37 | 14
  ICS | 30 | 15
  LAMA | 6 | 35
  SABA/SAMA | 9 | 22
  a-CHOL | 2 | 8
  LABA/LAMA | 0 | 9
  ICS/LABA/LAMA | 0 | 8
  PDE4 | 0 | 8
  a-IgE | 2 | 1
  LABA | 2 | 1
  IL-5 | 2 | 0

14. Primary Outcome: Number of Days in Hospital for Asthma and COPD
Description: The number of days for which the participant was hospitalized for asthma and COPD was summarized using data from EHR-based healthcare utilization
Time Frame: Up to 6 months
Population: All Enrolled Population
Measure: Number; unit: Days
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Days | 0 | 0

15. Primary Outcome: Number of Participants Who Received Short-acting Beta-agonist Therapy
Description: Participants who received SABA were summarized using data from EHR-based healthcare utilization.
Time Frame: Up to 6 months
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Participants | 85 | 85

16. Primary Outcome: Change From Baseline in COPD Assessment Test (CAT) Score-COPD Cohort Only
Description: The CAT is an 8 item questionnaire (cough, sputum, chest tightness, breathlessness, going up hills/stairs, activity limitation at home, confidence leaving the home, and sleep and energy) that measures health status of participants with COPD. Participants completed each question by rating their experience on a 6 point scale ranging from 0 (maximum impairment) to 5 (no impairment). Total score was calculated by summing the non-missing scores on the eight items and ranged from 0-40. Higher scores indicated greater disease impact. Week 1 was considered as Baseline. Change from Baseline was calculated as value at the specified time point minus Baseline value.
Time Frame: Baseline (Week 1) and Weeks 5, 9, 13, 17, 21 and 25
Population: All Enrolled Population. A total of 92 participants were included in the analysis; however, only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | COPD Cohort
Number analyzed (Participants) | 92
Scores on a scale
  Week 5, n=71: number analyzed (Participants) | 71
  Week 5, n=71 | 0 [-4 to 4]
  Week 9, n=67: number analyzed (Participants) | 67
  Week 9, n=67 | 0 [-3 to 3]
  Week 13, n=60: number analyzed (Participants) | 60
  Week 13, n=60 | 1 [-3 to 3]
  Week 17, n=56: number analyzed (Participants) | 56
  Week 17, n=56 | 0.5 [-3 to 4]
  Week 21, n=50: number analyzed (Participants) | 50
  Week 21, n=50 | 1.5 [-2 to 4]
  Week 25, n=48: number analyzed (Participants) | 48
  Week 25, n=48 | 0 [-3 to 4]

17. Primary Outcome: Change From Baseline in Asthma Control Test (ACT) Score-asthma Cohort Only
Description: The ACT is a validated self-administered questionnaire utilizing 5 questions to assess asthma control on a 5-point categorical scale (1 to 5). Total score was calculated as the sum of scores from 5 questions and ranged from 5 to 25. Higher scores indicated better control of asthma. Week 1 was considered as Baseline. Change from Baseline was calculated as value at the specified time point minus Baseline value.
Time Frame: Baseline (Week 1) and Weeks 5, 9, 13, 17, 21 and 25
Population: All Enrolled Population. A total of 95 participants were included in the analysis; however, only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Asthma Cohort
Number analyzed (Participants) | 95
Scores on a scale
  Week 5, n=72: number analyzed (Participants) | 72
  Week 5, n=72 | 0 [-1 to 2]
  Week 9, n=54: number analyzed (Participants) | 54
  Week 9, n=54 | 0 [-2 to 1]
  Week 13, n=62: number analyzed (Participants) | 62
  Week 13, n=62 | 0 [-1 to 2]
  Week 17, n=59: number analyzed (Participants) | 59
  Week 17, n=59 | 0 [-2 to 2]
  Week 21, n=47: number analyzed (Participants) | 47
  Week 21, n=47 | 0 [-1 to 2]
  Week 25, n=46: number analyzed (Participants) | 46
  Week 25, n=46 | 0 [-1 to 2]

18. Primary Outcome: Median Rescue Medication Use
Description: The use of rescue medication by participants were monitored by attaching a sensor to rescue inhaler.
Time Frame: Weeks 1, 5, 9, 13, 17, 21, 25
Population: All Enrolled Population. Only those participants with rescue medication sensors were analyzed.
Measure: Median (Inter-Quartile Range); unit: Occasions per day
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 69 | 76
Occasions per day
  Week 1 | 0.3 [0.1 to 1.3] | 0.6 [0.1 to 1.7]
  Week 5 | 0.2 [0 to 1] | 0.4 [0.1 to 1.3]
  Week 9 | 0.1 [0 to 0.6] | 0.3 [0 to 0.9]
  Week 13 | 0.1 [0 to 0.9] | 0.3 [0 to 0.9]
  Week 17 | 0 [0 to 0.5] | 0.3 [0 to 0.9]
  Week 21 | 0 [0 to 0.3] | 0.3 [0 to 0.7]
  Week 25 | 0 [0 to 0.3] | 0.3 [0 to 1]

19. Primary Outcome: Percentage of Participants With Maintenance Compliance
Description: The use of maintenance therapy by participants were monitored by attaching a sensor to maintenance inhaler.
Time Frame: Weeks 1, 5, 9, 13, 17, 21 and 25
Population: All Enrolled Population. Only those participants with maintenance medication sensors were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 71 | 59
Percentage of Participants
  Week 1 | 68 | 64
  Week 5 | 59 | 56
  Week 9 | 54 | 54
  Week 13 | 52 | 50
  Week 17 | 48 | 48
  Week 21 | 48 | 49
  Week 25 | 46 | 48

20. Primary Outcome: Number of Participants Who Completed Exit Interview
Description: An exit interview were conducted to obtain relevant feedback from participants regarding the study, study devices and electronic PRO platform. Exit surveys were triggered via the study-supplied iPad to each participant when they completed (or withdrew from) the study.
Time Frame: Up to 6 Months
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Cohort | COPD Cohort
Number analyzed (Participants) | 96 | 98
Participants | 96 | 80

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Adverse events (AEs) and serious adverse events (SAEs) were observed in All Enrolled Population.
Arm/Group | Asthma Cohort | COPD Cohort
All-Cause Mortality (participants affected / at risk) | 0/96 | 1/98
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/98
Other Adverse Events (participants affected / at risk) | 0/96 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03357341/Prot_SAP_000.pdf